CLINICAL TRIAL: NCT00131391
Title: A 2-Year Study (1-Year Weight Loss Followed by 1-Year Prevention of Weight Regain) to Assess the Safety, Tolerability and Efficacy of Taranabant (MK0364) in Obese Patients Followed by a 1-Year Extension
Brief Title: A Study of MK0364 in Obese Patients (0364-014)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The overall profile does not support development for obesity
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0364-014; 2005_034
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — N-(3-(4-chlorophenyl)-2-(3-cyanophenyl)-1-methylpropyl)-2-methyl-2-((5-(trifluoromethyl)pyridin-2-yl)oxy)propanamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Phase A/B; Arm 1 (Placebo Comparator): Phase A: Arm 1: MK0364 Pbo capsule once daily. Phase B: Patients who continue into Part B will remain in the same treatment arm they were assigned to in Part A and will receive the following: Arm 1: MK0364 Pbo capsule once daily.
  Interventions: Drug: Comparator: placebo
- Phase A/B: Arm 2 (Experimental): Phase A: Arm 2: MK0364 4 mg capsule once daily. Phase B: Patients who continue into Part B will remain in the same treatment arm they were assigned to in Part A and will receive the following: Arm 2: MK0364 4 mg capsule once daily.
  Interventions: Drug: Comparator: taranabant
- Phase A/B: Arm 3 (Experimental): Phase A: Arm 3: MK0364 6 mg capsule once daily. Phase B: Patients who continue into Part B will remain in the same treatment arm they were assigned to in Part A and will receive the following: Arm 3: MK0364 Pbo capsule once daily.
  Interventions: Drug: Comparator: taranabant; Drug: Comparator: placebo
- Phase A/B: Arm 4 (Experimental): Phase A: Arm 4: MK0364 6 mg capsule once daily. Phase B: Patients who continue into Part B will remain in the same treatment arm they were assigned to in Part A and will receive the following: Arm 4: MK0364 2 mg capsule once daily.
  Interventions: Drug: Comparator: taranabant
- Phase A/B: Arm 5 (Experimental): Phase A: Arm 5: MK0364 6 mg capsule once daily. Phase B: Patients who continue into Part B will remain in the same treatment arm they were assigned to in Part A and will receive the following: Arm 5: MK0364 4 mg capsule once daily.
  Interventions: Drug: Comparator: taranabant
- Phase A/B: Arm 6 (Experimental): Phase A: Arm 6: MK0364 6 mg once daily. Phase B: Patients who continue into Part B will remain in the same treatment arm they were assigned to in Part A and will receive the following: Arm 6: MK0364 6 mg capsule once daily.
  Interventions: Drug: Comparator: taranabant

INTERVENTIONS:
Drug: Comparator: taranabant — taranabant 2 mg capsule, 4 mg capsule, 6 mg capsule. 52 week treatment period.
  Other Names: MK0364
  Arms: Phase A/B: Arm 2; Phase A/B: Arm 3; Phase A/B: Arm 4; Phase A/B: Arm 5; Phase A/B: Arm 6
Drug: Comparator: placebo — Placebo capsule once daily . 52 week treatment period.
  Arms: Phase A/B: Arm 3; Phase A/B; Arm 1

SUMMARY:
A worldwide study in obese patients to assess the efficacy, safety, and tolerability of an investigational drug.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 30-43 kg/m2

Exclusion Criteria:

* History of major psychiatric disorder
* History of seizures or at high risk of developing seizures
* Blood pressure greater than 160/100
* Fasting blood glucose greater than 126 mg/dL
* Triglycerides greater than 600 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2005-07; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Decreases body weight; prevention of weight regain; safety and tolerability | 2 Years

SECONDARY OUTCOMES:
Decreases waist circumference, decreases the proportion of patients with metabolic syndrome, decreases triglycerides, decreases non-HDL-C, decreases LDL-C, decreases fasting insulin, decreases FPG; increases HDL-C, increases insulin sensitivity | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC